CLINICAL TRIAL: NCT07092930
Title: Evaluation of the Synergistic Effect of β-alanine and Sodium Bicarbonate Supplementation on Physical Capacity and Blood Biochemical Markers Concentrations in Trained Female Basketball Players
Brief Title: Effects of β-alanine and Sodium Bicarbonate Supplementation on Physical Capacity and Biochemical Markers Concentrations
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Poznan University of Physical Education (Other)
Responsible Party: Principal Investigator, Krzysztof Durkalec-Michalski, Prof., Poznan University of Physical Education
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZDS2025_0001
Record Dates: First submitted 2025-07-18; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Supplementation; Sports; Female Athletes
Keywords: Beta-alanine; Sodium bicarbonate; Ergogenic aids; Sports nutrition; Team sports; Physical capacity; Body composition; Blood and urine biochemical markers

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- BA and SB supplementation (first group) (Experimental)
  Interventions: Dietary Supplement: BA and SB supplementation
- BA and PL2 supplementation (second group) (Experimental)
  Interventions: Dietary Supplement: BA and PL2 supplementation
- PL1 and SB supplementation (third group) (Experimental)
  Interventions: Dietary Supplement: PL1 and SB supplementation
- PL1 and PL2 supplementation (fourth group) (Placebo Comparator)
  Interventions: Dietary Supplement: PL1 and PL2 supplementation

INTERVENTIONS:
Dietary Supplement: BA and SB supplementation — Assigned Interventions:
  * Beta-alanine (BA)
  * Sodium bicarbonate (SB)
  Description:
  • Participants receive beta-alanine and sodium bicarbonate
  Intervention list & supplementation details:
  1. Beta-alanine (BA)
     * Form: Gelatin capsules
     * Substance: Pure beta-alanine
     * Daily dose: 6.4 g/day
     * Dosing schedule: Four equal servings taken with meals (breakfast, lunch, snack, dinner)
     * Supplementation period: days 1 to 28
  2. Sodium bicarbonate (SB)
     * Form: Gelatin capsules
     * Substance: Pure sodium bicarbonate
     * Daily dose: 0.3 g/kg body mass per day
     * Dosing schedule: Three equal servings taken with meals (breakfast, lunch, dinner)
     * Supplementation period: days 21 to 28 of BA or PL1 supplementation
  Rationale:
  • This group tests the combined effects of BA and SB
  Arms: BA and SB supplementation (first group)
Dietary Supplement: BA and PL2 supplementation — Participants in this intervention group will undergo chronic supplementation with beta-alanine (BA) and an inert placebo (PL2) matched to the sodium bicarbonate (SB) protocol.
  * Beta-alanine (pure, in gelatin capsules) will be administered at a total daily dose of 6.4 g, divided into four servings taken with meals, over a period of 28 consecutive days.
  * PL2 (placebo matched to SB, in gelatin capsules) will be administered from Day 21 to Day 28 of beta-alanine supplementation, at a daily dose of 0.3 g per kg of body mass, divided into three equal servings taken with meals.
  This group allows for evaluation of the isolated effects of BA supplementation when combined with a placebo comparator to SB
  Arms: BA and PL2 supplementation (second group)
Dietary Supplement: PL1 and SB supplementation — Assigned Interventions:
  * Placebo matched to BA (PL1)
  * Sodium bicarbonate (SB)
  Description:
  • Participants receive only sodium bicarbonate as the active compound and placebo capsules matching the BA protocol.
  Intervention list & supplementation details:
  1. Placebo matched to BA (PL1)
     * Form: Gelatin capsules
     * Substance: Inert substance matched in appearance and dosing schedule to BA
     * Daily dose: 6.4 g/day
     * Dosing schedule: Four equal servings taken with meals (breakfast, lunch, snack, dinner)
     * Supplementation period: days 1 to 28
  2. Sodium bicarbonate (SB)
     * Form: Gelatin capsules
     * Substance: Pure sodium bicarbonate
     * Daily dose: 0.3 g/kg body mass per day
     * Dosing schedule: Three equal servings taken with meals (breakfast, lunch, dinner)
     * Supplementation period: days 21 to 28 of BA or PL1 supplementation
  Rationale:
  • This group tests the isolated effects of SB
  Arms: PL1 and SB supplementation (third group)
Dietary Supplement: PL1 and PL2 supplementation — Assigned Interventions:
  * Placebo matched to BA (PL1)
  * Placebo matched to SB (PL2)
  Description:
  • Participants receive two matched placebos.
  Intervention list & supplementation details:
  1. Placebo matched to BA (PL1)
     * Form: Gelatin capsules
     * Substance: Inert substance matched in appearance and dosing schedule to BA
     * Daily dose: 6.4 g/day
     * Dosing schedule: Four equal servings taken with meals (breakfast, lunch, snack, dinner)
     * Supplementation period: days 1 to 28
  2. Placebo matched to SB (PL2)
     * Form: Gelatin capsules
     * Substance: Inert substance matched in appearance and timing to SB
     * Daily dose: 0.3 g/kg body mass per day
     * Dosing schedule: Three equal servings taken with meals (breakfast, lunch, dinner)
     * Supplementation period: days 21 to 28 of BA or PL1 supplementation
  Rationale:
  • This serves as the control group for comparison with all active intervention arms.
  Arms: PL1 and PL2 supplementation (fourth group)

SUMMARY:
This randomized, double-blind, placebo-controlled, parallel-group study aims to evaluate the potential synergistic effect of beta-alanine (BA) and sodium bicarbonate (SB) supplementation, compared to their separate administration or placebo (PL), on physical performance and selected blood biochemical markers in highly trained female basketball players.

DETAILED DESCRIPTION:
Beta-alanine (BA) and sodium bicarbonate (SB) are commonly proposed as ergogenic aids due to their potential to enhance intracellular (BA) and extracellular (SB) buffering capacities, thereby improving physical performance. However, there is a lack of evidence regarding their potential synergistic effects, particularly in female athletes. Existing studies have primarily focused on male participants, despite emerging evidence suggesting sex-specific physiological responses to supplementation. Furthermore, research shows that females exhibit a high willingness to participate in scientific studies, underlining the importance of including female cohorts in sports supplementation research. To date, no randomized, double-blind, placebo-controlled trials have examined the combined and separate effects of BA and SB using a four-arm design (BA+SB, BA+PL2, PL1+SB, PL1+ PL2). Only one study to date has focused on chronic SB supplementation, whereas the majority have used acute protocols. Additionally, there is a notable lack of data on the use of BA and SB in team sports such as basketball, where repeated high-intensity efforts are dominant. Therefore, this study aims to investigate the chronic effects of BA and SB supplementation (administered individually or in combination) on physical capacity and selected blood biochemical markers in highly trained female basketball players, using a randomized, double-blind, placebo-controlled, parallel-group design.

ELIGIBILITY:
Inclusion Criteria:

* written consent to participate,
* general good health condition,
* a current medical clearance to practice sports,
* training experience: at least 4 years,
* minimum of 4 workout sessions (in the discipline covered by the study) a week.

Exclusion Criteria:

* current injury,
* any health-related contraindication,
* declared general feeling of being unwell,
* taking supplements, especially ergogenic supplements that modulate extra- and intracellular capacity 3 months prior to research (except taking protein and/or carbohydrate powders, isotonic drinks),
* unwilling to follow the study protocol.

Ages: 16 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Changes in anaerobic capacity during Wingate Anaerobic Test (WAnT) | During the first study visit on the first day and during the second study visit after 28 days of intervention.
  Assessment of peak power (PP), average power (AP), minimum power (MP), power drop (PD) [W (Watts)] using the Monark 894E ergometer (measured before and after incremental cycling test (ICT)) before and after supplementation (BA - beta-alanine; SB - sodium bicarbonate; PL - placebo; with BA+SB, BA+PL2, PL1+SB, or PL1+PL2).
Changes in Countermovement Jump (CMJ) performance | During the first study visit on the first day and during the second study visit after 28 days of intervention.
  Assessment of three consecutive countermovement jump (CMJ) heights [cm (centimetres)] using the Microgate system, measured at rest and after the entire exercise procedure, both before and after supplementation.
Changes in aerobic capacity during incremental cycling test (ICT) | During the first study visit on the first day and during the second study visit after 28 days of intervention.
  Assessment of time to exhaustion [s (seconds)] during an incremental cycling test (ICT) using Ergoline E100P-K, measured before and after supplementation (with BA+SB, BA+PL2, PL1+SB, or PL1+PL2).
Changes in blood bicarbonate, base excess, anion gap, and lactate concentrations | During the first study visit on the first day and during the second study visit after 28 days of intervention.
  Assessment of bicarbonate, base excess, anion gap, lactate [mmol/L] measured in capillary blood at rest, after warm-up, and after the entire exercise procedure, before and after supplementation (with BA+SB, BA+PL2, PL1+SB, or PL1+PL2).
Changes in hydrogen ion concentration | During the first study visit on the first day and during the second study visit after 28 days of intervention.
  Assessment of hydrogen ion concentration [nmol/L] measured in capillary blood at rest, after warm-up, and after the entire exercise procedure, before and after supplementation (with BA+SB, BA+PL2, PL1+SB, or PL1+PL2).

SECONDARY OUTCOMES:
Analysis of dietary energy intake | 48 h before the first study visit and the second study visit after 28 days of intervention.
  Assessment of energy intake [kcal (kilocalories)], before and after supplementation (with BA+SB, BA+PL2, PL1+SB, or PL1+PL2).
Analysis of dietary macronutrient intake | 48 h before the first study visit and the second study visit after 28 days of intervention.
  Assessment of macronutrients intake (proteins, carbohydrates, fats) [g (grams)], before and after supplementation (with BA+SB, BA+PL2, PL1+SB, or PL1+PL2).
Changes in rate of perceived exertion | During the first study visit on the first day and during the second study visit after 28 days of intervention.
  The Borg RPE Scale ranges from 6 (no exertion at all) to 20 (maximal exertion). Higher scores indicate greater subjective perceived physical effort. The scale will be administered in accordance with the original methodology described by Borg (1982).
Changes in heart rate | During the first study visit on the first day and during the second study visit after 28 days of intervention.
  Assessment of heart rate (HR) [bpm (beats per minute)] during the entire exercise procedure, measured before and after supplementation (with BA+SB, BA+PL2, PL1+SB, or PL1+PL2).
Changes in gastrointestinal symptoms | During the first study visit on the first day and during the second study visit after 28 days of intervention.
  Assessment of gastrointestinal (GI) symptoms using the adapted and validated Gastrointestinal and Related Complaints Questionnaire, via a self-reported symptom severity scale [0-10], administered at rest and after the exercise procedure, before and after supplementation (with BA+SB, BA+PL2, PL1+SB, or PL1+PL2).
  The questionnaire assesses 19 symptoms: stomach problems, nausea, dizziness, headache, flatulence, urge to urinate, urge to defecate, belching, heartburn, bloating, stomach cramps, intestinal cramps, urge to vomit, vomiting, diarrhoea, left side ache, right side ache, muscle cramps, and cold shivering.
  Each symptom is rated from 0 (no symptoms) to 10 (severe symptoms). Higher scores indicate greater gastrointestinal symptom severity. The scale will be administered in accordance with the methodology described by Jeukendrup et al. (2000).
Changes in body mass, fat-free mass and fat mass | During the first study visit on the first day and during the second study visit after 28 days of intervention.
  Assessment of body mass, fat-free mass and fat mass [kg (kilograms)] at rest, before and after supplementation (with BA+SB, BA+PL2, PL1+SB, or PL1+PL2).
Changes in total body water content | During the first study visit on the first day and during the second study visit after 28 days of intervention.
  Assessment of total body water, extracellular and intracellular water [% (percentage)] at rest, before and after supplementation (with BA+SB, BA+PL2, PL1+SB, or PL1+PL2).
Changes in lymphocytes, monocytes, granulocytes, red blood cells and platelets | During the first study visit on the first day and during the second study visit after 28 days of intervention.
  Assessment of blood cells (WBC), lymphocytes (LYM), monocytes (MON), granulocytes (GRA), red blood cells (RBC) and platelets (PLT) [count/L] will be performed in capillary blood collected at rest, after warm-up, and after the entire exercise procedure, before and after supplementation (with BA+SB, BA+PL2, PL1+SB, or PL1+PL2).
Changes in platelets distribution width and platelets large cell ratio | During the first study visit on the first day and during the second study visit after 28 days of intervention.
  Assessment of platelets distribution width (PDW) and platelets large cell ratio (PLCR) [%] will be performed in capillary blood collected at rest, after warm-up, and after the entire exercise procedure, before and after supplementation (with BA+SB, BA+PL2, PL1+SB, or PL1+PL2).
Changes in hemoglobin and mean corpuscular hemoglobin concentration | During the first study visit on the first day and during the second study visit after 28 days of intervention.
  Assessment of hemoglobin and mean corpuscular hemoglobin concentration [mmol/L] will be performed in capillary blood collected at rest, after warm-up, and after the entire exercise procedure, before and after supplementation (with BA+SB, BA+PL2, PL1+SB, or PL1+PL2).
Changes in hematocrit | During the first study visit on the first day and during the second study visit after 28 days of intervention.
  Assessment of hematocrit (HCT) [L/L] will be performed in capillary blood collected at rest, after warm-up, and after the entire exercise procedure, before and after supplementation (with BA+SB, BA+PL2, PL1+SB, or PL1+PL2).
Changes in mean corpuscular volume, mean platelet volume, red blood cell distribution width | During the first study visit on the first day and during the second study visit after 28 days of intervention.
  Assessment of hematological markers [fL] will be performed in capillary blood collected at rest, after warm-up, and after the entire exercise procedure, before and after supplementation. The analysis will include mean corpuscular volume (MCV), mean platelet volume (MPV), read blood cell distribution width (RDW) [fL], before and after supplementation (with BA+SB, BA+PL2, PL1+SB, or PL1+PL2).
Changes in mean corpuscular hemoglobin | During the first study visit on the first day and during the second study visit after 28 days of intervention.
  Assessment of mean corpuscular hemoglobin (MCH) [fmol] will be performed in capillary blood collected at rest, after warm-up, and after the entire exercise procedure, before and after supplementation (with BA+SB, BA+PL2, PL1+SB, or PL1+PL2).
Changes in alanine aminotransferase, aspartate aminotransferase, creatine kinase and lactate dehydrogenase | During the first study visit on the first day and during the second study visit after 28 days of intervention.
  Assessment of alanine aminotransferase (ALAT), aspartate aminotransferase (ASAT), creatine kinase (CK) and lactate dehydrogenase (LDH) [U/L] will be performed in capillary blood collected at rest, after warm-up, and after the entire exercise procedure, before and after supplementation (with BA+SB, BA+PL2, PL1+SB, or PL1+PL2).
Changes in urea and magnesium | During the first study visit on the first day and during the second study visit after 28 days of intervention.
  Assessment of urea and magnesium (Mg) [mmol/L] will be performed in capillary blood collected at rest, after warm-up, and after the entire exercise procedure, before and after supplementation (with BA+SB, BA+PL2, PL1+SB, or PL1+PL2).
Changes in creatinine | During the first study visit on the first day and during the second study visit after 28 days of intervention.
  Assessment of creatinine concentration [μmol/L] will be performed in capillary blood collected at rest, after warm-up, and after the entire exercise procedure, before and after supplementation (with BA+SB, BA+PL2, PL1+SB, or PL1+PL2).
Changes in iron and unsaturated iron binding capacity | During the first study visit on the first day and during the second study visit after 28 days of intervention.
  Assessment of iron and unsaturated iron binding capacity (UIBC) [μg/dL] will be performed in capillary blood collected at rest, after warm-up, and after the entire exercise procedure, before and after supplementation (with BA+SB, BA+PL2, PL1+SB, or PL1+PL2)
Changes in transferrin | During the first study visit on the first day and during the second study visit after 28 days of intervention.
  Assessment of transferrin [g/L] will be performed in capillary blood collected at rest, after warm-up, and after the entire exercise procedure, before and after supplementation (with BA+SB, BA+PL2, PL1+SB, or PL1+PL2).
Changes in ferritin | During the first study visit on the first day and during the second study visit after 28 days of intervention.
  Assessment of ferritin [μg/mL] will be performed in capillary blood collected at rest, after warm-up, and after the entire exercise procedure, before and after supplementation (with BA+SB, BA+PL2, PL1+SB, or PL1+PL2).
Changes in potassium, sodium, ionized calcium, chloride, osmolality | During the first study visit on the first day and during the second study visit after 28 days of intervention.
  Assessment of potassium (cK⁺), sodium (cNa⁺), ionized calcium (cCa²⁺), chloride (cCl-), osmolality (mOsm.c) [mmol/L] measured in capillary blood at rest, after warm-up, and after the entire exercise procedure, before and after supplementation (with BA+SB, BA+PL2, PL1+SB, or PL1+PL2).
Changes in urine specific gravity | During the first study visit on the first day and during the second study visit after 28 days of intervention.
  Assessment of urine specific gravity (USG) measured in urine at rest, before and after supplementation (with BA+SB, BA+PL2, PL1+SB, or PL1+PL
Changes in protein, glucose, ketones, urobilinogen, bilirubin | During the first study visit on the first day and during the second study visit after 28 days of intervention.
  Assessment of protein (PRO), glucose (GLU), ketones (KET), urobilinogen (UBG), bilirubin (BIL) [mg/dL] measured in urine at rest, before and after supplementation (with BA+SB, BA+PL2, PL1+SB, or PL1+PL2).
Changes in pH | During the first study visit on the first day and during the second study visit after 28 days of intervention.
  Assessment of pH measured in urine at rest, before and after supplementation (with BA+SB, BA+PL2, PL1+SB, or PL1+PL2).
Changes in urine erythrocytes and leukocytes | During the first study visit on the first day and during the second study visit after 28 days of intervention.
  Assessment of erythrocytes (BLD), leukocytes (LEU) [cells/μL] measured in urine at rest, before and after supplementation (with BA+SB, BA+PL2, PL1+SB, or PL1+PL2).
Changes in urine luteinizing hormone and nitrite | During the first study visit on the first day and during the second study visit after 28 days of intervention.
  Assessment of luteinizing hormone (LH) and nitrite (NIT) [positive/negative] measured in urine at rest, before and after supplementation (with BA+SB, BA+PL2, PL1+SB, or PL1+PL2).

CONTACTS AND LOCATIONS:
Overall Officials: Krzysztof Durkalec-Michalski, PhD, Study Chair — Department of Sports Dietetics, Poznan University of Physical Education Poznań
Locations (1):
- Department of Sports Dietetics, Poznan University of Physical Education Poznań, Poznan, Wielkopolska, Poland

IPD SHARING:
Plan to Share IPD: Yes
Shared data will be exclusively related to the level of recorded indicators, without personal data. The data obtained will be attached to scientific publications, depending on the requirements of the journal.
  De-identified individual participant data (IPD), including timepoint-specific values of primary and secondary outcome measures (e.g., performance results, hematological and physiological parameters), will be shared. Data will be made available upon reasonable request to qualified researchers for non-commercial academic purposes, following publication of the primary results. Requests should be directed to the corresponding author via institutional email. A data use agreement may be required.

REFERENCES:
- [Background] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893
- [Background] Jeukendrup AE, Vet-Joop K, Sturk A, Stegen JH, Senden J, Saris WH, Wagenmakers AJ. Relationship between gastro-intestinal complaints and endotoxaemia, cytokine release and the acute-phase reaction during and after a long-distance triathlon in highly trained men. Clin Sci (Lond). 2000 Jan;98(1):47-55. PMID 10600658